CLINICAL TRIAL: NCT03136367
Title: Comparative Effectiveness of Encounter Decision Aids for Early-Stage Breast Cancer Across Socioeconomic Strata
Brief Title: What Matters Most: Choosing the Right Breast Cancer Surgery for You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Washington University School of Medicine (Other); Montefiore Medical Center (Other); NYU Langone Health (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Marie-Anne Durand, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D17063
Record Dates: First submitted 2017-04-25; First posted 2017-05-02 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: encounter decision aids; shared decision making; socioeconomic status; disparities; decision quality
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Three-arm randomized controlled superiority trial with stratification by SES and randomization at the clinician level. Patient enrollment will occur at five cancer centers in the United States. Patients will be enrolled in one of the three arms based on the clinician they are seeing as a part of their care.
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blinded to the clinician randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Option Grid (Experimental): Patients in this arm will receive the Option Grid for breast cancer surgery, an encounter decision aid, when they first meet with the breast surgeon to discuss their surgical options for breast cancer treatment.
  Interventions: Other: Option Grid
- Arm 2: Picture Option Grid (Experimental): Patients in this arm will receive the Picture Option Grid for breast cancer surgery, an encounter decision aid, when they first meet with the breast surgeon to discuss their surgical options for breast cancer treatment.
  Interventions: Other: Picture Option Grid
- Arm 3: Usual Care (No Intervention): In the usual care arm, surgeons provided their standard information about breast cancer

INTERVENTIONS:
Other: Option Grid — The Option Grid(TM) encounter decision aid for early stage breast cancer surgery is a one-page, evidence-based summary of available options presented in a tabular format.
  Other Names: Option Grid for Breast Cancer Surgery; Breast cancer: surgical options
  Arms: Arm 1: Option Grid
Other: Picture Option Grid — The Picture Option Grid was derived from the Option Grid for early stage breast cancer. It uses the same evidence and integrates images and simpler text, thus exploiting pictorial superiority. The Picture Option Grid has been specifically designed for women of lower SES and low health literacy.
  Other Names: Early-stage breast cancer: What's right for me?
  Arms: Arm 2: Picture Option Grid

SUMMARY:
What Matters Most is a study that aims to determine how best to help women of lower socioeconomic status make high-quality decisions about early stage breast cancer treatments. What Matters Most will be comparing two decision aids used in the clinic visit to usual care (what normally happens in the clinic). The first decision aid (Option Grid) presents evidence-based information about lumpectomy and mastectomy in a tabular format using text only. The second decision aid (Picture Option Grid) presents evidence-based information about lumpectomy and mastectomy using pictures, pictographs and simplified text. What Matters Most aims to show that the interventions can reduce disparities in decision-making and treatment choice between women of high and low SES.

DETAILED DESCRIPTION:
Background and Significance

Breast cancer is the most commonly diagnosed malignancy in women. Despite improvements in survival, women of low socioeconomic status (SES) diagnosed with early stage breast cancer:

* Continue to experience poorer doctor-patient communication, lower satisfaction with surgery and decision making, and higher decision regret compared to women of higher SES;
* Often play a passive role in decision making;
* Are less likely to undergo breast-conserving surgery (BCS);
* Are less likely to receive optimal care.

Those differences are disparities that predominantly affect women of low SES with early stage breast cancer, irrespective of race or ethnicity. For early stage breast cancer, low SES is a stronger predictor of poorer outcomes, treatment received and death, than race or ethnicity. The investigators define low SES as a lower income, lower educational attainment, and uninsured or state-insured status

Although BCS is the recommended treatment for early stage breast cancer (stages I to IIIA), research confirms equivalent survival between mastectomy and BCS. Both options are offered yet have distinct harms and benefits, valued differently by patients. The patient and stakeholder partners involved in this study have emphasized the critical importance of supporting women in making high quality breast cancer surgery decisions (good knowledge and alignment between the patient's choice, values and priorities) irrespective of SES and health literacy. Yet, research shows that women of low SES are not usually involved in an informed, patient-centered dialogue about surgery choice. There is no evidence that women of low SES have distinct preferences that explain a lower uptake of BCS and limited engagement in decision making. Further, communication strategies are not typically adapted to women of low SES and low health literacy. Most decision aids for breast cancer have been designed for highly literate audiences, with poor accessibility and readability. Simpler, shorter decision aids delivered in the clinical encounter (encounter decision aids) may be more beneficial to underserved patients, and could reduce disparities. It is critical to determine how to effectively support women of low SES in making informed breast cancer surgery choices.

Study Aims

First, the investigators will assess the comparative effectiveness of two effective encounter decision aids (Option Grid and Picture Option Grid) against usual care on decision quality (primary outcome), shared decision making, treatment choice and other secondary outcomes across socioeconomic strata (Aim 1). Second, the investigators aim to explore the effect of the Picture Option Grid on disparities in decision making (decision quality, knowledge, and shared decision making), treatment choice, as well as mediation and moderation effects (Aim 2). Third, in order to maximize the implementation potential, the investigators will explore strategies that promote the encounter decision aids' sustained use and dissemination using a theoretical implementation model (Aim 3).

Study Description

The investigators will conduct a three-arm, multi-site randomized controlled superiority trial with stratification by SES (Aims 1 and 2) and randomization at the clinician level. One thousand, one hundred patients (half of higher SES and half of lower SES) will be recruited from five large cancer centers. In preparation for the trial (Year 01), the investigators will conduct semi-structured interviews with women of low SES who have completed treatment for early stage breast cancer to adapt the "What Matters Most to You" subscale of the Decision Quality Instrument (DQI) for women of low SES. Lastly, the investigators will use interviews, field-notes, and observations to explore strategies that promote the interventions' sustained use and dissemination using the Normalization Process Theory (Aim 3). Community-Based Participatory Research will be used throughout the trial (with continuous patient and stakeholder involvement).

Women 18 years and older with a confirmed diagnosis of early stage breast cancer (I to IIIA) from both higher and lower SES will be included in the trial, provided they have a basic command of English, Spanish, or Mandarin. About 367 patients will be recruited per arm.

Both interventions have been developed, tested, and shown to be effective. The Option Grid (intervention 1) is a one-page evidence-based summary of available options presented in a tabular format, listing the trade-offs that patients normally consider when making breast cancer surgery decisions. The Picture Option Grid (intervention 2) uses the same evidence and tabular layout, but it is tailored to women of lower SES and low health literacy and includes simple text and images. Because decision aids are not routinely available in real world settings, usual care is a coherent and legitimate comparator. It will include the provision of usual information resources about breast cancer but will exclude the provision of other decision aids.

Secondary outcome measures will include treatment choice, the validated 3-item CollaboRATE measure of shared decision-making (SDM), Chew's validated one-item health literacy screening question, PROMIS, an 8-item validated anxiety short form, EQ-5D-5L, a validated, standardized 6-item quality of life measure, and four items from COST, a validated financial toxicity measure. Participants will also be asked to estimate their out-of-pocket expenses over the past month. All measures will be available in English, Spanish, and Mandarin. Observer OPTION5 will be used to rate the level of shared decision making in the clinical encounter.

A regression framework (logistic regression, linear regression, mixed effect regression models, generalized estimating equations) and mediation analyses will be used in the analysis. The investigators will also use multiple informants analysis to measure and examine SES and multiple imputation to manage missing data. Heterogeneity of treatment effects analyses for SES, age, ethnicity, race, literacy, language, and study site will be performed. The investigators will also use the recordings of surgical consultations to analyze the conversations about costs and treatment recommendations made by providers.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth;
* 18 years and older;
* Confirmed diagnosis (via biopsy) of early stage breast cancer (stages I-IIIA);
* Eligible for both breast-conserving surgery and mastectomy based on medical records and clinician's opinion before surgery;
* Spoken English, Spanish, or Mandarin Chinese.

Exclusion Criteria:

* Transgender men and women;
* Women who have undergone prophylactic mastectomy;
* Women with visual impairment;
* Women with a diagnosis of severe mental illness or severe dementia;
* Women with inflammatory breast carcinoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In order to be in this trial, participants must have been assigned female at birth. Transgender men will also be excluded as their treatment course would be managed on a case-by-case basis.
Enrollment: 571 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ann Durand, MSc, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (5):
- United States (5):
  - Washington University in St. Louis, St Louis, Missouri
  - Norris Cotton Cancer Center, Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CN, Wetschler MH, Chang Y, Belkora JK, Moy B, Partridge A, Sepucha KR. Measuring decision quality: psychometric evaluation of a new instrument for breast cancer chemotherapy. BMC Med Inform Decis Mak. 2014 Aug 20;14:73. doi: 10.1186/1472-6947-14-73. PMID 25142035
- [Background] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Barr PJ, O'Malley AJ, Tsulukidze M, Gionfriddo MR, Montori V, Elwyn G. The psychometric properties of Observer OPTION(5), an observer measure of shared decision making. Patient Educ Couns. 2015 Aug;98(8):970-6. doi: 10.1016/j.pec.2015.04.010. Epub 2015 Apr 29. PMID 25956069
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Elwyn G, Thompson R, John R, Grande SW. Developing IntegRATE: a fast and frugal patient-reported measure of integration in health care delivery. Int J Integr Care. 2015 Mar 27;15:e008. doi: 10.5334/ijic.1597. eCollection 2015 Jan-Mar. PMID 26034467
- [Background] Pickard AS, De Leon MC, Kohlmann T, Cella D, Rosenbloom S. Psychometric comparison of the standard EQ-5D to a 5 level version in cancer patients. Med Care. 2007 Mar;45(3):259-63. doi: 10.1097/01.mlr.0000254515.63841.81. PMID 17304084
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Sepucha KR, Belkora JK, Chang Y, Cosenza C, Levin CA, Moy B, Partridge A, Lee CN. Measuring decision quality: psychometric evaluation of a new instrument for breast cancer surgery. BMC Med Inform Decis Mak. 2012 Jun 8;12:51. doi: 10.1186/1472-6947-12-51. PMID 22681763
- [Derived] Schubbe D, Yen RW, Saunders CH, Elwyn G, Forcino RC, O'Malley AJ, Politi MC, Margenthaler J, Volk RJ, Sepucha K, Ozanne E, Percac-Lima S, Bradley A, Goodwin C, van den Muijsenbergh M, Aarts JWM, Scalia P, Durand MA. Implementation and sustainability factors of two early-stage breast cancer conversation aids in diverse practices. Implement Sci. 2021 May 10;16(1):51. doi: 10.1186/s13012-021-01115-1. PMID 33971913
- [Derived] Durand MA, Yen RW, O'Malley AJ, Schubbe D, Politi MC, Saunders CH, Dhage S, Rosenkranz K, Margenthaler J, Tosteson ANA, Crayton E, Jackson S, Bradley A, Walling L, Marx CM, Volk RJ, Sepucha K, Ozanne E, Percac-Lima S, Bergin E, Goodwin C, Miller C, Harris C, Barth RJ Jr, Aft R, Feldman S, Cyr AE, Angeles CV, Jiang S, Elwyn G. What matters most: Randomized controlled trial of breast cancer surgery conversation aids across socioeconomic strata. Cancer. 2021 Feb 1;127(3):422-436. doi: 10.1002/cncr.33248. Epub 2020 Nov 10. PMID 33170506
- [Derived] Durand MA, Yen RW, O'Malley AJ, Politi MC, Dhage S, Rosenkranz K, Weichman K, Margenthaler J, Tosteson ANA, Crayton E, Jackson S, Bradley A, Volk RJ, Sepucha K, Ozanne E, Percac-Lima S, Song J, Acosta J, Mir N, Elwyn G. What matters most: protocol for a randomized controlled trial of breast cancer surgery encounter decision aids across socioeconomic strata. BMC Public Health. 2018 Feb 13;18(1):241. doi: 10.1186/s12889-018-5109-2. PMID 29439691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2017 and February 2019, we screened 2,057 of a target 2,200 patients; 1,031 patients remained eligible. We approached 885 eligible patients, of which 622 (76.6%) consented. Sixteen surgeons saw 571 of 622 consented patients.
Pre-assignment Details: Sixteen surgeons saw 571 of 622 consented patients. The imbalanced allocation to arms was due to differences in the number of patients seen by each surgeon, or changes in their role or attendance. Of 440 patients who consented to recording, we collected 311 (70.7%) usable recordings.
Period: T1 Consultation
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Started | 66 | 248 | 257
Completed | 64 (received the intervention) | 241 | 256
Not Completed | 2 | 7 | 1
Not completed — discontinued mistakenly included | 2 | 6 | 1
Not completed — Discontinued other | 0 | 1 | 0
Period: T2 Post-consultation
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Started | 64 | 241 | 256
Completed | 61 | 235 | 225
Not Completed | 3 | 6 | 31
Not completed — Withdrawal by Subject | 1 | 1 | 5
Not completed — discontinued mistakenly included | 2 | 2 | 17
Not completed — Discontinued other | 0 | 2 | 6
Not completed — Discontinued transferred care | 0 | 0 | 3
Not completed — Discontinued lost contact | 0 | 1 | 0
Period: T3 1 Week After Surgery
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Started | 61 | 235 | 225
Completed | 51 | 203 | 194
Not Completed | 10 | 32 | 31
Not completed — Discontinued mistakenly included | 5 | 9 | 8
Not completed — Discontinued transferred care | 2 | 11 | 14
Not completed — other discontinued | 2 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 6 | 2
Not completed — Discontinued lost contact | 1 | 2 | 4
Period: T4 12 Weeks After Surgery
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Started | 51 | 203 | 194
Completed | 49 | 198 | 185
Not Completed | 2 | 5 | 9
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Death | 0 | 1 | 3
Not completed — discontinued lost contact | 1 | 0 | 0
Not completed — discontinued transferred care | 0 | 1 | 5
Not completed — discontinued mistakenly included | 0 | 0 | 1
Period: T5 1 Year After Surgery
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Started | 49 | 198 | 185
Completed | 13 | 62 | 56
Not Completed | 36 | 136 | 129
Not completed — discontinued mistakenly included | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Discontinued lost contact | 1 | 6 | 0
Not completed — Lost to Follow-up | 2 | 22 | 15
Not completed — study ended before due | 31 | 103 | 110
Not completed — logistical issues prevented contact | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: 622 participants consented to take part but 6 participants withdrew consent immediately before or during baseline, leaving 616 participant with baseline information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care | Total
Number analyzed (Participants) | 69 | 276 | 271 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.5) | 58.9 (13.0) | 60.4 (12.2) | 59.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 276 | 271 | 616
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 13 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 37 | 40 | 96
  White | 46 | 218 | 208 | 472
  More than one race | 1 | 4 | 8 | 13
  Unknown or Not Reported | 1 | 4 | 11 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Decision Quality: Knowledge Subscale
Description: Change in decision quality, measured using the validated 16-item Decision Quality Worksheet for Breast Cancer Surgery. Decision quality is measured through three constructs: knowledge, decision process, and concordance. Knowledge is five questions that results in a score from 0 to 5 with higher numbers indicating higher knowledge. Decision process is a measure how much shared decision making process occurred, based on patient-report. It is a seven-item scale with higher numbers indicating higher shared decision process. For the concordance score, patients rated their goals and concerns on an 11-point importance scale from 0 (not important at all) to 10 (extremely important). They also indicated which surgery they intended to have at T2. A concordance summary score (0-100%) indicated the percentage of patients who received a treatment that matched their stated preference.
Time Frame: Immediately before the index surgical consultation visit, immediately after the index surgical consultation visit and at one week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  Immediately before the index surgical consultation visit | 2.83 (1.29) | 2.95 (1.22) | 2.77 (1.21)
  Immediately after the index surgical consultation visit | 2.82 (1.13) | 2.90 (1.07) | 2.74 (1.07)
  One week post-surgery | 3.00 (1.11) | 2.88 (1.05) | 2.87 (1.12)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.045, Mixed Models Analysis — Adjusted for repeated within-patient measurements; Mixed effects linear regression that accounted for clinician and site clustering and was adjusted for surgeon and patient characteristics
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.20, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.82, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Change in Decision Quality: Decison Process Subscale
Description: Change in decision quality, measured using the validated 16-item Decision Quality Worksheet for Breast Cancer Surgery. Decision quality is measured through three constructs: knowledge, decision process, and concordance. Knowledge is five questions that results in a score from 0 to 5 with higher numbers indicating higher knowledge. Decision process is a measure how much shared decision making process occurred, based on patient-report. It is a seven-item scale from 0 to 7 with higher numbers indicating higher shared decision process. For the concordance score, patients rated their goals and concerns on an 11-point importance scale from 0 (not important at all) to 10 (extremely important). They also indicated which surgery they intended to have at T2. A concordance score indicated the percentage of patients who received a treatment that matched their stated preference.
Time Frame: Immediately after the index surgical consultation visit and at one week post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  Immediately after the index surgical consultation visit | 5.66 (1.24) | 5.47 (1.58) | 4.57 (2.10)
  One week post-surgery | 5.67 (1.26) | 5.02 (1.73) | 4.64 (1.95)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.048, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.015, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.43, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Change in Decision Quality: Concordance Subscale
Description: Change in decision quality, measured using the validated 16-item Decision Quality Worksheet for Breast Cancer Surgery. Decision quality is measured through three constructs: knowledge, decision process, and concordance. Knowledge is five questions that results in a score from 0 to 5 with higher numbers indicating higher knowledge. Decision process is a measure how much shared decision making process occurred, based on patient-report. It is a seven-item scale with higher numbers indicating higher shared decision process. For the concordance score, patients rated their goals and concerns on an 11-point importance scale from 0 (not important at all) to 10 (extremely important). They also indicated which surgery they intended to have at T2. A concordance summary score (0-100%) indicated the percentage of patients who received a treatment that matched their stated preference at T2 (lumpectomy vs mastectomy).
Time Frame: Immediately after the index surgical consultation visit and at one week post-surgery
Population: Only participants who remained in the trial through when they had their surgery were analyzed for this outcome in order to assess the match between treatment intent and treatment received.
Measure: Number; unit: percentage with treatment match
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 43 | 148 | 168
percentage with treatment match | 95.3 | 92.9 | 95.4
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mixed effects linear regression that accounted clustering and was adjusted for surgeon and patient characteristics
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.34, Mixed Models Analysis; Mixed effects linear regression that accounted clustering and was adjusted for surgeon and patient characteristics
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.165, Mixed Models Analysis; Mixed effects linear regression that accounted clustering and was adjusted for surgeon and patient characteristics

4. Secondary Outcome: Number of Participants Who Chose Lumpectomy or Mastectomy as Their Treatment Choice
Description: Treatment choice, or which surgical or treatment option the patient chose, mastectomy or lumpectomy (breast conserving surgery)
Time Frame: 1 week post-surgery
Population: The number of participants analyzed for treatment choice was different from other outcome measures as it is based on the number of participants for whom treatment choice data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 52 | 200 | 192
Participants
  lumpectomy | 42 | 161 | 146
  mastectomy | 10 | 39 | 46

5. Secondary Outcome: Change in Quality of Life
Description: Quality of life reported by the patient measured using the validated 6-item EQ-5D-5L measure. We used the available resources from EuroQol to convert EQ-5D-5L states into an index value, using the EQ-5D-5L crosswalk value sets. Index values ranged from full health (1) and to no health (-0.109), according to the US crosswalk value set.
Time Frame: Immediately before the index surgical consultation visit and at 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  Immediately before the index surgical consultation visit | 0.83 (0.13) | 0.82 (0.13) | 0.82 (0.14)
  12 weeks post-surgery | 0.82 (0.10) | 0.85 (0.13) | 0.82 (0.12)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.25, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.89, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.54, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Anxiety
Description: Patient-reported anxiety, measured using the validated 8-item PROMIS anxiety short form. Each question was coded from one to five. Total scores were obtained by scoring the raw score of each item answered. The lowest possible raw score was 8; the highest possible raw score was 40 with higher numbers indicating higher anxiety.
Time Frame: Immediately before the index surgical consultation visit, immediately after the index surgical consultation visit, at 1 week post-surgery, and at 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  Immediately before the index surgical consultation visit | 20.8 (6.8) | 20.2 (7.4) | 20.7 (7.7)
  immediately after the index surgical consultation visit | 20.0 (6.7) | 20.4 (8.1) | 20.6 (7.9)
  1 week post-surgery | 17.2 (7.3) | 17.0 (7.1) | 17.1 (6.7)
  12 weeks post-surgery | 13.1 (6.5) | 13.0 (5.6) | 14.9 (6.9)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.72, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.41, McNemar — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.28, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Shared Decision-making (Self-reported)
Description: Self-reported shared decision-making about breast cancer surgical options measured using the validated 3-item CollaboRATE measure. Each item was rated on a scale from 0 to 9 with a possible score range from 0 to 27. We dichotomized this measure using the top score approach, grouping participants scoring 9 on all three items versus all others.
Time Frame: Immediately after the index surgical consultation visit
Measure: Number (95% Confidence Interval); unit: percentage of patients with a top score
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
percentage of patients with a top score | 73 [48 to 99] | 76 [55 to 97] | 58 [52 to 65]
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.12, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.78, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Shared Decision-making (Observed)
Description: Shared decision-making observed during the surgical consultation, measured using the validated observer-rated OPTION5. The five items on the measure ask raters to score the consultation on how much the clinician: 1) confirms that alternatives exist, 2) reassures that they will support the patient to become informed, 3) gives information or checks understanding about the options, 4) makes an effort to elicit the patient's preferences, and 5) integrates the patient's elicited preferences. Each of the five items is scored from zero to four for a summary score ranging from zero to 20 and a scaled score ranging from zero to 100. Higher numbers indicate more shared decision making was observed.
Time Frame: During the index surgical consultation visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 41 | 143 | 127
score on a scale | 69.92 [42.51 to 95.16] | 65.72 [41.84 to 89.45] | 41.02 [36.20 to 45.85]
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p < 0.01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Decision Regret
Description: Patient-reported feelings of decision regret, measured using the validated 5-item decision regret scale. Items 2 and 4 were reverse coded so a higher number indicated more regret. Scores were then converted to a 0-100 scale by subtracting 1 from each item then multiply by 25. To obtain a final score, the items were summed and averaged. A score of 0 meant no regret and a score of 100 meant high regret.
Time Frame: At 1 week post-surgery, 12 weeks post-surgery, and 1 year post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  1 week post-surgery | 10.9 (13.9) | 8.1 (12.3) | 12.9 (14.5)
  12 weeks post-surgery | 12.0 (15.9) | 7.6 (12.3) | 10.8 (16.2)
  1 year post-surgery | 10.4 (14.1) | 6.0 (10.3) | 7.6 (14.3)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.06, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.65, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.36, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Integration of Health Care Delivery
Description: Patient-reported measure of integration of healthcare delivery, measured using IntegRATE, a 4-item scale. IntegRATE sum scores are determined by summing each participant's scores across the 4 items (range 0-12). A higher score indicates higher integration.
Time Frame: Immediately before the index surgical consultation visit and at 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
Number analyzed (Participants) | 66 | 248 | 257
score on a scale
  Immediately before the index surgical consultation visit | 10.4 (1.8) | 10.2 (2.0) | 10.3 (1.9)
  12 weeks post-surgery | 10.9 (1.1) | 10.8 (1.5) | 10.6 (1.8)
Statistical Analysis 1: Comparison: Arm 2: Picture Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.11, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm 1: Option Grid vs Arm 3: Usual Care; Test type: Superiority; p = 0.037, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Arm 1: Option Grid vs Arm 2: Picture Option Grid; Test type: Superiority; p = 0.28, Mixed Models Analysis — Adjusted for repeated within-patient measurements; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Exploration of Strategies That Promote the Interventions' Sustained Use and Dissemination
Description: Semi-structured interviews with clinic stakeholders and patients 12 weeks post-surgery, field notes, and clinic observations to explore strategies that promote the interventions' sustained use and dissemination
Time Frame: 12 weeks post-surgery (patients) or after trial participation ended (surgeons)
Population: The results are reported in two groups: patients and all surgeons. The data collection method used was semi-structured interview (using a purposive sampling technique). This was a qualitative exploration of the data. We did not interview all participants but only purposively selected 42 participants in the intervention arms. Some results in this section only apply to patients (e.g., helped with decision) and some only apply to surgeons (e.g., would recommend to other health professionals).
Measure: Count of Participants; unit: Participants
Groups:
- Patients in Intervention Arms: Patients in this group received either the Option Grid or Picture Option Grid as a part of their care. Only patients in the intervention arms were interviewed for this outcome measure.
- Surgeons Involved in the Trial: This group included all surgeons who participated in the trial. All surgeons were interviewed for this outcome measure.
Arm/Group | Patients in Intervention Arms | Surgeons Involved in the Trial
Number analyzed (Participants) | 42 | 16
Participants
  Patients: number analyzed (Participants) | 42 | 0
  Patients: Aid affected treatment decision | 30 |
  Patients: Aid was part of normal routine | 29 |
  Patients: Want paper-based materials | 40 |
  Patients: Thought receiving aid from the surgeon is best | 30 |
  Patients: Open to receiving the aid in virtual formats | 30 |
  Patients: Open to receiving/giving aid before appointment | 15 |
  Patients: Aid would be helpful for lower literacy patients | NA — This category/result only applies to surgeons. |
  Patients: Recommended other health professionals use the aid | NA — This category/result only applies to surgeons. |
  Patients: Were able to integrate the aid into their routine | NA — This category/result only applies to surgeons. |
  All trial surgeons: number analyzed (Participants) | 0 | 16
  All trial surgeons: Aid affected treatment decision |  | NA — This category/result only applies to patients.
  All trial surgeons: Aid was part of normal routine |  | NA — This category/result only applies to patients.
  All trial surgeons: Want paper-based materials |  | NA — This category/result only applies to patients.
  All trial surgeons: Thought receiving aid from the surgeon is best |  | NA — This category/result only applies to patients.
  All trial surgeons: Open to receiving the aid in virtual formats |  | NA — This category/result only applies to patients.
  All trial surgeons: Open to receiving/giving aid before appointment |  | 8
  All trial surgeons: Aid would be helpful for lower literacy patients |  | NA — This category/result only applies to surgeons in the intervention arms.
  All trial surgeons: Recommended other health professionals use the aid |  | 16
  All trial surgeons: Were able to integrate the aid into their routine |  | NA — This category/result only applies to surgeons in the intervention arms.
  Intervention surgeons: number analyzed (Participants) | 0 | 11
  Intervention surgeons: Aid affected treatment decision |  | NA — This category/result only applies to patients.
  Intervention surgeons: Aid was part of normal routine |  | NA — This category/result only applies to patients.
  Intervention surgeons: Want paper-based materials |  | NA — This category/result only applies to patients.
  Intervention surgeons: Thought receiving aid from the surgeon is best |  | NA — This category/result only applies to patients.
  Intervention surgeons: Open to receiving the aid in virtual formats |  | NA — This category/result only applies to patients.
  Intervention surgeons: Open to receiving/giving aid before appointment |  | NA — This category/result only applies to patients or the entire surgeon group analysis.
  Intervention surgeons: Aid would be helpful for lower literacy patients |  | 6
  Intervention surgeons: Recommended other health professionals use the aid |  | NA — This category/result only applies to patients or the entire surgeon group analysis.
  Intervention surgeons: Were able to integrate the aid into their routine |  | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm 1: Option Grid | Arm 2: Picture Option Grid | Arm 3: Usual Care
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/248 | 4/257
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/248 | 0/257
Other Adverse Events (participants affected / at risk) | 0/66 | 0/248 | 0/257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT03136367/Prot_SAP_ICF_000.pdf